CLINICAL TRIAL: NCT03539952
Title: CHELATE STUDY: Trientine Tetrahydrochloride (TETA 4HCL) for the Treatment of Wilson's Disease
Brief Title: Trientine Tetrahydrochloride (TETA 4HCL) for the Treatment of Wilson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Orphalan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMPO-131-002
Record Dates: First submitted 2018-05-04; First posted 2018-05-30 (Actual); Results first posted 2023-04-20 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Wilson Disease
MeSH Terms: conditions — Hepatolenticular Degeneration | interventions — Penicillamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Penicillamine arm (Active Comparator): Patients randomized to penicillamine during the postrandomisation and 1st extension period
  Interventions: Drug: Penicillamine (D1-W12); Drug: Penicillamine (W12-W60); Drug: TETA 4HCL (60-<W108)
- Trientine arm (Experimental): Patients randomized to TETA 4HCl during the postrandomisation and 1st extension period
  Interventions: Drug: Penicillamine (D1-W12); Drug: TETA 4HCL (W12-60); Drug: TETA 4HCL (60-<W108)

INTERVENTIONS:
Drug: Penicillamine (D1-W12) — Penicillamine during baseline period (D1-W12)
  Other Names: D-penicillamine
Drug: TETA 4HCL (W12-60) — TETA 4HCL during post randomisation and 1st extension period (W12-W60)
  Other Names: trientine tetrahydrochloride
  Arms: Trientine arm
Drug: Penicillamine (W12-W60) — Penicillamine during rondomisation and 1st extension period period (W12-W60)
  Other Names: D-Penicillamine
  Arms: Penicillamine arm
Drug: TETA 4HCL (60-<W108) — TETA 4HCL during 2nd extension period (W60-<W108)
  Other Names: trientine tetrahydrochloride

SUMMARY:
This is a multicenter, randomized, open-label study with an active standard-of-care comparator (penicillamine)

DETAILED DESCRIPTION:
This is a multicenter, randomized, open label study with an active standard-of-care comparator.

Stable patients who are already considered to be stable on their standard-of-care penicillamine chelation therapy for at least 1 year will enroll in the study and enter a 12-week Penicillamine Baseline Period comprising of 1 month (4 weeks) run-in period followed by a 2 month (8 weeks) evaluation period. During this time all patients will continue to take their current penicillamine under study conditions. At the end of the Penicillamine Baseline Period, patients who fulfill the protocol definition of being adequately controlled and tolerating penicillamine will be randomized in a 1:1 ratio to receive either TETA 4HCl or to continue to receive penicillamine. There is then a 24-week Post-randomization Phase comprising of a 1 month (4 weeks) run-in period for both treatment arms and a 5 month (20 weeks) evaluation period.

Patients who successfully complete the 24-week Post-randomization Phase of the study will have the opportunity to enter an Extension Phase. In the first version of the clinical trial protocol, the intention was to have an 18 month (72 weeks) Extension Phase. During the first 24 weeks of the Extension Phase, subjects would continue receiving their allocated TETA 4HCl or penicillamine (i.e., up to Week 60 of the study). Thereafter all patients were receiving TETA 4HCl for a further 48 weeks (i.e., from Week 60 to Week 108). Study clinic visits occur were scheduled every 6 months in the Extension Phase.

With the final version of the protocol, the Extension Phase stopped at Week 60. Patients who already passed the Week 60 visit were allowed to end the study at the next planned visit.

As a consequece end of treatment varied Week 60 and Week 108

ELIGIBILITY:
Inclusion Criteria:

1. Patient is able to provide, and has provided, written informed consent
2. Written documentation has been obtained in accordance with the relevant country and local privacy requirements, where applicable, including: For US sites: Authorization for Use and Release of Health Research Study Information and for EU sites: Data Protection Consent
3. Male or female, aged ≥ 18 and ≤ 75 years of age at time of consent
4. Patient has a diagnosis of Wilson's disease, as defined by a prior or current Leipzig score of ≥ 4
5. Patient's Wilson's disease is clinically stable, in the opinion of the investigator, and being treated with penicillamine for at least 1 year (52 weeks) prior to the screening/enrolment visit
6. Patient is on a stable dose and regimen of penicillamine for at least 4 months (16 weeks) prior to the screening/enrolment visit (other prescribed treatments for Wilson's disease not permitted during this study)
7. No anticipated need that patient will require additional pharmacological therapies other than study medication, including prescribed zinc therapy, for the management of copper levels during the study
8. Patient must be willing to maintain stable diet throughout the study, and avoid foods with high copper content, including the Penicillamine Baseline Period
9. Patient considered suitable to receive therapy with both TETA 4HCl and penicillamine administered twice a day
10. Negative central laboratory tests for HIV and viral hepatitis (results will be available after start of run-in period)
11. For female patients of childbearing potential, negative urine pregnancy test (at screening/enrolment visit and prior to randomization)
12. For females of childbearing potential, use of a reliable form of contraceptive
13. Patient is considered as able to complete study requirements and attend the study visits, in the opinion of the investigator

    Additional inclusion criteria following receipt of Screening laboratory results
14. Patient is adequately controlled and tolerating penicillamine therapy as defined by fulfilment of all of the following: a. Serum non-ceruloplasmin bound copper (NCC) level between ≥ 25 and ≤ 150 μg/L* b. 24-hour urinary copper excretion of between ≥ 100 and ≤ 900 μg/24 hours* c. Alanine transaminase (ALT) < 2 times upper limit of normal* d. No other laboratory or clinical findings that would prevent continuation of maintenance therapy, in the opinion of the investigator

    * Based on results from screening/enrolment visit samples for which can be taken within ± 7 days of visit. Result should be within the assay limits of quantification for the sample. The ranges in μmol of copper are 0.40 to 2.38 μmol/L for NCC and 1.59 to 14.29 for 24-hour urinary copper excretion (using division by 63 of value in μg per Walshe, 2011). In the event that one or more of the above lab values fall outside the specified range, it can be repeated, including at the Week 4 and Week 8 visits.

    Additional inclusion criteria at Week 12 visit (end of Penicillamine Baseline Period) and prior to randomization
15. Patient is adequately controlled and tolerating penicillamine therapy as defined by fulfilment of all of the following criteria:

    1. Serum non-ceruloplasmin bound copper (NCC) level between ≥ 25 and ≤ 150 μg/L*
    2. 24-hour urinary copper excretion of between ≥ 100 and ≤ 900 μg/24 hours**
    3. Alanine transaminase (ALT) < 2 times upper limit of normal*
    4. No other laboratory or clinical findings that would prevent continuation of maintenance therapy, in the opinion of the investigator

       * Based on lab values from Week 8 visit; ** Based on lab value from Week 4 visit as routinely not performed at Week 8 visit, however can also be based on value at Week 8 visit if a repeat (unscheduled) urinary copper excretion was performed at this visit. Result should be within the assay limits of quantification for the sample. The ranges in μmol of copper are 0.40 to 2.38 μmol/L for NCC and 1.59 to 14.29 for 24-hour urinary copper excretion (using division by 63 of value in μg per Walshe, 2011). In the event that one or more of the above lab values fall outside the specified range, it can be repeated. The repeat value(s) must be available prior to randomization at Week 12 and, if within specified range, the patient can continue to randomization. If a patient fails this additional criterion at the end of the Penicillamine Baseline Period, the patient can return to the start of the run-in period i.e. Day 1 (but only once). A negative urinary pregnancy test is also required prior to randomization for females of childbearing potential.

Exclusion Criteria:

1. Patient is in 'de-coppering' phase of treatment for Wilson's disease, in the opinion of the investigator
2. Patient evidence of uncontrolled liver disease, including but not limited to:

   1. Modified Nazer score of > 4 (result may not be available until after start of run in period since based on lab results*)
   2. decompensated cirrhosis
   3. acute hemolytic anemia
   4. acute hepatitis
   5. hepatic malignancy
   6. evidence of acute liver failure
3. Cause of patient's liver disease is due to another condition, in the investigator's opinion
4. Patient has severe anemia defined as hemoglobin of ≤ 9 g/dL (result will be available after start of run-in period*)
5. Patient has experienced a gastrointestinal bleed within 6 months (24 weeks) prior to screening/enrolment visit
6. Patient has renal impairment defined as creatinine clearance of ≤ 30 mL/min (result may not be available until after start of run-in period*), or patient has nephritis or nephrotic syndrome, in the opinion of the investigator
7. Patient has neurological disease that prevents swallowing of study medication (e.g., requires a nasogastric feeding tube) or requires intensive in-patient medical care
8. Patient is currently taking medication containing trientine for management of Wilson's disease or has taken it within 4 months (16 weeks) of screening/enrolment visit
9. Patient is currently receiving prescribed zinc therapy for management of Wilson's disease or has taken it within 4 months (16 weeks) of screening/enrolment visit
10. Patient is taking any of the following concomitant therapies: gold therapy, antimalarial therapy, cytotoxic drugs, oxyphenbutazone, phenyl butazone
11. Patient has a known intolerance, allergy or sensitivity to penicillamine (that is uncontrolled) or to TETA 4HCl, including any component of the study medication
12. For female patients of childbearing potential, planning a pregnancy during study period or currently nursing
13. For female patients of childbearing potential, unable or unwilling to use a reliable form of contraceptive throughout the study
14. Patient is currently participating in another therapeutic study, or has previously participated in a therapeutic study within 30 days of screening/enrolment visit (or longer, if local requirements specify this)
15. Patient has any condition or in any situation which, in the investigator's opinion, puts the patient at significant risk, could confound study results, or may interfere significantly with the patient's participation in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2020-08-19 (Actual); Study Completion 2022-01-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- Yale University School of Medicine, New Haven, Connecticut, United States
- KU Leuven, Department of Clinical and Experimental Medicine, Leuven, Belgium
- Brazil (3):
  - Hospital Nossa Senhora das Graças (HNSG), Curitiba
  - Nucleo de Pesquisa e Desenvolvimento de Medicamentos - Universidade Federal do Ceará - Rodolfo Teófilo, Fortaleza
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo
- Hepato-gastroenterologisk afd, Aarhus, Denmark
- France (2):
  - Hospital mother children, Bron
  - Centre National de Référence Wilson, Hôpital Lariboisière, Paris
- Germany (2):
  - Innere Medizin, Heidelberg
  - Poliklinik Hepatologie/Transplantationsambulanz, Munich
- Italy (2):
  - A.O. San Paolo Milano, Milan
  - DiSCOG Gastroenterology Unit, Padua
- Institute of Psychiatry and Neurology, Warsaw, Poland
- United Kingdom (2):
  - University of Surrey, Department of Clinical and Experimental Medicine, Guildford, Surrey
  - Leeds Teaching Hospitals NHS Trust, Leeds

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schilsky ML, Czlonkowska A, Zuin M, Cassiman D, Twardowschy C, Poujois A, Gondim FAA, Denk G, Cury RG, Ott P, Moore J, Ala A, D'Inca R, Couchonnal-Bedoya E, D'Hollander K, Dubois N, Kamlin COF, Weiss KH; CHELATE trial investigators. Trientine tetrahydrochloride versus penicillamine for maintenance therapy in Wilson disease (CHELATE): a randomised, open-label, non-inferiority, phase 3 trial. Lancet Gastroenterol Hepatol. 2022 Dec;7(12):1092-1102. doi: 10.1016/S2468-1253(22)00270-9. Epub 2022 Sep 30. PMID 36183738
- [Derived] Ott P, Sandahl T, Ala A, Cassiman D, Couchonnal-Bedoya E, Cury RG, Czlonkowska A, Denk G, D'Inca R, de Assis Aquino Gondim F, Moore J, Poujois A, Twardowschy CA, Weiss KH, Zuin M, Kamlin COF, Schilsky ML. Non-ceruloplasmin copper and urinary copper in clinically stable Wilson disease: Alignment with recommended targets. JHEP Rep. 2024 May 6;6(8):101115. doi: 10.1016/j.jhepr.2024.101115. eCollection 2024 Aug. PMID 39139457

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was enrolled on 03 September 2018, the last patient completed the Week 36 visit (for primary analysis) on 19 August 2020, and the last patient visit in the study was on 18 January 2022.
Pre-assignment Details: After enrolment, patients entered a 12-week run-in period. This is referred to the Penicillamine Baseline Period. During this time, all patients received penicillamine, allowing dose adjustments to reach clinical and laboratory stability criteria. At the end of this 12-week period, patients were randomized 1:1 ratio to either continue penicillamine or receive TETA 4HCl if protocol definition of stability were met in addition to an independent assessment from a panel of WD specialists.
Groups:
- Penicillamine: Male and female clinically stable Wilson Disease patients, aged ≥18 and ≤75, receiving penicillamine treatment for at least 1 year, stable dose for at least 4 months prior to enrolment. Patients continued on their current penicillamine therapy from week 1 till 12, the baseline period. When confirmed stable, patients were randomized to continue penicillamine (control) treatment for the 24 weeks post-randomization phase (week 12-36). Patients completing the 24-weeks post-randomization phase, were offered to enter a 24 week extension period on their allocated (control) Penicillamine. At the end of the extension period (study end), all patients were offered continuing involvement by switching to TETA 4HCl.
- TETA 4HCl: Male and female clinically stable Wilson Disease patients, aged ≥18 and ≤75, receiving penicillamine treatment for at least 1 year, stable dose for at least 4 months prior to enrolment. Patients continued on their current penicillamine therapy from week 1 till 12, the baseline period. When confirmed stable, patients were randomized to open label TETA 4HCl (intervention) treatment for the 24 weeks post-randomization phase (week 12-36). Patients completing the 24-weeks post-randomization phase, were offered to enter a 24 week extension period on their allocated (intervention) TETA 4HCl. At the end of the extension period (study end), all patients were offered continuing involvement by switching to or continuing TETA 4HCl.
Period: Penicillamine Baseline Period (Day1-W12)
Arm/Group | Penicillamine | TETA 4HCl
Started | 77 | 0
Completed | 53 | 0
Not Completed | 24 | 0
Not completed — Baseline run-in failure | 24 | 0
Period: Post-randomization Period (Week 12-36)
Arm/Group | Penicillamine | TETA 4HCl
Started (The number of participants starting the Post-randomization period in one of the two arms is equal to the number of subjects that completed the baseline period, i.e. before randomisation) | 27 (Patients completing period 1 and randomized to receive penicillamine) | 26 (Patients completing period 1 and randomized to receive TETA 4HCl)
Completed | 26 | 26
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Extension Post Random. (Week 36-60)
Arm/Group | Penicillamine | TETA 4HCl
Started | 26 | 26
Completed | 19 | 23
Not Completed | 7 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Not further documented | 3 | 1
Period: All on TETA 4HCl, From wk 60 Till 108max
Arm/Group | Penicillamine | TETA 4HCl
Started | 19 | 23
Completed | 19 | 21
Not Completed | 0 | 2
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Penicillamine Arm: Comparator: Penicillamine
  TETA 4HCL: TETA 4HCL
  Penicillamine: Penicillamine
- TETA 4HCL Arm: Active Treatment
  TETA 4HCL: TETA 4HCL
  Penicillamine: Penicillamine
- Total: Total of all reporting groups
Arm/Group | Penicillamine Arm | TETA 4HCL Arm | Total
Number analyzed (Participants) | 27 | 26 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 25 | 51
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (13.43) | 42.0 (15.63) | 43.6 (14.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 12 | 28
  Male | 11 | 14 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 24 | 21 | 45
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 2 | 3 | 5
  United States | 1 | 1 | 2
  Brazil | 6 | 4 | 10
  Denmark | 1 | 1 | 2
  Poland | 4 | 4 | 8
  Italy | 2 | 3 | 5
  United Kingdom | 1 | 2 | 3
  France | 2 | 2 | 4
  Germany | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Serum NCC Concentration
Description: The primary outcome of efficacy was serum NCC by speciation assay (μg/L), with comparative analysis of mean difference between the two groups 24 weeks after randomization. The non-inferiority margin was set at -50 μg/L.
Time Frame: Week 36
Population: ITT
Measure: Mean (Standard Error); unit: µg/L
Arm/Group | Penicillamine Arm | TETA 4HCL Arm
Number analyzed (Participants) | 25 | 26
µg/L | 46.5 (5.69) | 58.7 (5.54)
Statistical Analysis 1: Comparison: Penicillamine Arm vs TETA 4HCL Arm; The primary endpoint was the assessment of the non-inferiority of TETA 4HCl in relation to D-penicillamine. The non-inferiority assessment was made on the basis of the mean serum NCC level at Week 36; Test type: Non-Inferiority — The primary efficacy analysis utilized the serum NCC values from all study visits that were analyzed using a restricted maximum likelihood based general linear model for correlated data. The correlation due to repeated measures was modeled by specifying the variance covariance matrix. Considering a comparison of means in both treatment arms (D-penicillamine minus TETA 4HCl) at the 1-sided 2.5% level of Type 1 error, a non-inferiority margin of 50 μg/L was used; Mean Difference (Final Values) = -9.2, Standard Error of Mean 7.49

2. Secondary Outcome: 24-hour Urinary Copper Excretion (UCE)
Description: 24-hour urinary copper excretion (μg/ 24 hr) from urine collected by the patient over a 24-hour period.
Time Frame: Week 36
Measure: Mean (Standard Error); unit: μg/24 hours
Groups:
- TETA 4HCL: Active Treatment
  TETA 4HCL: TETA 4HCL
  Penicillamine: Penicillamine
- Penicillamine: Comparator: Penicillamine
  TETA 4HCL: TETA 4HCL
  Penicillamine: Penicillamine
Arm/Group | TETA 4HCL | Penicillamine
Number analyzed (Participants) | 26 | 27
μg/24 hours | 274.5 (45.59) | 510.8 (47.77)

3. Secondary Outcome: Clinical Global Impression of Change (CGIC) Rating Scale
Description: The clinician will rate the change in the patient's Wilson's disease relative to the prior study clinic visit using a 7-point scale to a specific statement: 'Please rate the change in the overall severity of the patients Wilson's disease compared to the previous study clinic visit".
  Available options were (1) very much improved; (2) much improved; (3) minimally improved; (4) no change; (5) minimally worse; (6), much worse; or (7) very much worse.
Time Frame: Week 36
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Penicillamine: Comparator:
  Penicillamine
- TETA 4HCL: Active Treatment
  TETA 4HCL
Arm/Group | Penicillamine | TETA 4HCL
Number analyzed (Participants) | 21 | 22
score on a scale | 4.1 (0.10) | 3.9 (0.05)

ADVERSE EVENTS:
Time Frame: From Day 1 up to Week 108 / End of Treatment
Description: Displayed (serious) adverse events were collected on randomized patients only. Note that treatment changed from one period to the next, depending on the period and the randomly assigned treatment arm.
  Patients randomized to the penicillamine arm received resp. Penicillamine, Penicillamine, Penicillamine and TETA 4HCl, from period 1 to 4.
  Whereas patients randomized to the TETA 4HCl arm received resp. Penicillamine, TETA 4HCl, TETA 4HCl and TETA 4HCl from period 1 to 4.
Groups:
- D1-W12 Penicillamine Arm; D1-W12 TETA 4HCl Arm: Penicillamine Baseline Period from Day 1 until randomization at W12
  In this period all patients received Penicillamine
- W12-W36 Penicllamine Arm: Post randomization phase, W12 until W36
  In this period all patients received their allocated treatement, i.e., Penicillamine
- W12-W36 TETA4HCl Arm: Post randomization phase, W12 until W36
  In this period all patients received their allocated treatement, i.e., TETA4HCl
- W36-60 Pencillamine Arm: Extension phase, W36 until W60
  In this period all patients received their allocated treatement, i.e., Penicillamine
- W36-60 TETA4HCl Arm: Extension phase, W36 until W60
  In this period all patients received their allocated treatement, i.e., TETA4HCl
- W60-108 Pencillamine Arm; W60-108 TETA4HCl Arm: Extension phase, W60 until <W108
  In this period all patients received TETA4HCL
Arm/Group | D1-W12 Penicillamine Arm | D1-W12 TETA 4HCl Arm | W12-W36 Penicllamine Arm | W12-W36 TETA4HCl Arm | W36-60 Pencillamine Arm | W36-60 TETA4HCl Arm | W60-108 Pencillamine Arm | W60-108 TETA4HCl Arm
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/26 | 0/27 | 0/26 | 0/26 | 0/26 | 0/19 | 1/23
Serious Adverse Events (participants affected / at risk) | 1/27 | 1/26 | 3/27 | 0/26 | 0/26 | 0/26 | 0/19 | 3/23
Other Adverse Events (participants affected / at risk) | 11/27 | 10/26 | 10/27 | 13/26 | 3/26 | 3/26 | 6/19 | 5/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D1-W12 Penicillamine Arm (N=27) | D1-W12 TETA 4HCl Arm (N=26) | W12-W36 Penicllamine Arm (N=27) | W12-W36 TETA4HCl Arm (N=26) | W36-60 Pencillamine Arm (N=26) | W36-60 TETA4HCl Arm (N=26) | W60-108 Pencillamine Arm (N=19) | W60-108 TETA4HCl Arm (N=23)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — SUSPICION OF DYSPLASTIC CHANGES IN LIVER CIRRHOTIC TISSUE IN LIVER MAGNETIC RESONANCE EXAMINATION
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Escherichia sepsis
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Escherichia sepsis
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — ARTERIOSCLEROSIS OF THE CONORARY ARTERY
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Cystitis
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Atrial fibrillation
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D1-W12 Penicillamine Arm (N=27) | D1-W12 TETA 4HCl Arm (N=26) | W12-W36 Penicllamine Arm (N=27) | W12-W36 TETA4HCl Arm (N=26) | W36-60 Pencillamine Arm (N=26) | W36-60 TETA4HCl Arm (N=26) | W60-108 Pencillamine Arm (N=19) | W60-108 TETA4HCl Arm (N=23)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (12) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (4) | 2 (4) | 5 (8) | 2 (4) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Mood swings (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-05-27): https://cdn.clinicaltrials.gov/large-docs/52/NCT03539952/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-18): https://cdn.clinicaltrials.gov/large-docs/52/NCT03539952/SAP_001.pdf